CLINICAL TRIAL: NCT07166003
Title: Effects of Neoadjuvant Immunotherapy on Patients With Lung Cancer: a Prospective, Observational Study
Brief Title: Efficacy of Neoadjuvant Immunotherapy in Patients With Lung Cancer
Acronym: NeoIP-Lung
Status: Recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 2025040620521402
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer, Non-Small Cell; Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pneumonectomy; Anterior Temporal Lobectomy; Radiotherapy; Antineoplastic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery: Patients will undergo surgery after neoadjuvant immunotherapy.
  Interventions: Procedure: Pneumonectomy; Procedure: lobectomy
- Non-surgery: Patients will receive non-surgical treatment after neoadjuvant treatment.
  Interventions: Radiation: radiotherapy; Drug: Anti-Tumor Drugs

INTERVENTIONS:
Procedure: Pneumonectomy — Patients will receive pneumonectomy after neoadjuvant treatment
  Groups: Surgery
Procedure: lobectomy — Patients will receive lobectomy after neoadjuvant immunotherapy.
  Groups: Surgery
Radiation: radiotherapy — Patients will receive radiotherapy after neoadjuvant immunotherapy.
  Groups: Non-surgery
Drug: Anti-Tumor Drugs — Patients will receive anti-tumor drugs.
  Groups: Non-surgery

SUMMARY:
The goal of this observational study is to learn about the long-term effects of neoadjuvant immunotherapy in patients with lung cancer. The main questions it aims to answer are:

* Does pneumonectomy bring more benefits for pateints than lobectomy?
* Does surgery bring more benefits for patients than non-surgery modalities (such as radiotherapy) after neoadjuvnat immunotherapy? Participants will receive neoadjuvant treatment and the study will analyze the data.

DETAILED DESCRIPTION:
This observational study aims to comprehensively evaluate the effectiveness and long-term clinical outcomes of neoadjuvant treatment in patients with lung cancer. Central to this investigation are two key questions: ·Does pneumonectomy bring more benefits for pateints than lobectomy?

* Does surgery bring more benefits for patients than non-surgery modalities (such as radiotherapy) after neoadjuvnat immunotherapy? Participants will receive neoadjuvant treatment, and through rigorous analysis of data, this study endeavors to provide nuanced insights into these fundamental queries, fostering advancements in clinical decision-making and patient management strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 79 years;
2. Received at least two cycles of neoadjuvant immunotherapy;
3. ECOG performance status score of 0;
4. Complete clinical information including imaging data available.

Exclusion Criteria:

1. Diagnosed with or suspected active autoimmune diseases;
2. Presence of EGFR/ALK sensitive mutations;
3. Pregnant or breastfeeding women;
4. Previous anti-tumor therapies including chemotherapy or radiotherapy;
5. History of organ transplantation or hematopoietic stem cell transplantation;
6. Interstitial pneumonia, pulmonary fibrosis, or severe emphysema;
7. Uncontrolled diabetes mellitus;
8. Uncontrolled hypertension.

Ages: 18 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with lung cancer who receive neoadjuvant immunotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2030-04-14 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | Event-free survival was defined as the time from neoadjuvant treatment to metastasis or death by any cause in the absence of metastasis, up to approximately 10 years.

SECONDARY OUTCOMES:
Overall survival | From date of neoadjuvant treatment until date of death due to any cause, up to approximately 10 years.
Perioperative Complication rate | Within 6 months after neoadjuvant treatment.
  Complications after the neoadjuvant treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, China